CLINICAL TRIAL: NCT01527981
Title: CBT for Adherence and Depression in Type 1 Diabetes
Brief Title: Cognitive Behavioral Therapy (CBT) for Adherence and Depression in Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven A. Safren, Director, Behavioral Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MGHBMED2172010
Record Dates: First submitted 2012-01-31; First posted 2012-02-07 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Depression; Type 1 Diabetes
Keywords: Depression; Diabetes; Adherence; Medication; Glucose; Insulin
MeSH Terms: conditions — Depression; Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- CBT-AD (Experimental): Participants received weekly one-hour CBT-AD sessions focusing on diabetes self-care and depression for approximately 10 sessions. Participants also had meetings with a registered dietitian and a nurse educator, focusing on nutritional management of diabetes and diabetes self-care education, respectively.
  Interventions: Behavioral: Cognitive behavioral therapy for adherence and depression

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for adherence and depression — Cognitive-behavioral therapy for adherence and depression (CBT-AD) is a weekly, psychosocial treatment focusing on depression and patients' adherence to diabetes self-care. Treatment consists of weekly one-hour sessions for approximately 10 sessions.
  Other Names: CBT-AD

SUMMARY:
This study is a pilot behavioral intervention trial, designed to initially examine cognitive behavioral therapy for medical adherence and depression (CBT-AD) in patients with depression and poorly controlled type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes that is poorly controlled (HbA1C greater than or equal to 8.0%) despite treatment with insulin.
* Diagnosis of major depression and/or dysthymia, or current subclinical symptoms of depression in spite of being treated with antidepressants.
* Age 18-80.
* If on an antidepressant, stable for two months. Oral hypoglycemic medications stable for 2 months, and insulin prescription stable for 2 months (if prescribed).

Exclusion Criteria:

* Active or untreated major mental illness that would interfere with participation (e.g., untreated psychosis), untreated/unstable bipolar disorder, eating disorder, mental retardation, dementia, or active suicidality.
* Unable or unwilling to provide informed consent.
* History of or current CBT for depression.
* Currently on dialysis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Changes in glucose monitoring | Baseline assessment; 4, 8, and 12 months post-intervention assessments
  We used electronic glucometers to measure participants' adherence to prescribed glucose self-monitoring, which record each time glucose was measured and the glucose level of each measurement.
Changes in insulin adherence | Baseline assessment; 4, 8, and 12 months post-intervention assessments
  We assessed adherence to participants' self-administered insulin through a self-report questionnaire.
Changes in depression severity | Baseline assessment; 4, 8, and 12 months post-intervention assessments
  Participants' depression severity was measured by clinician-administered measures (Montgomery-Asberg Depression Rating Scale) and self-report measures (Center for Epidemiological Studies Depression Scale). Clinician-delivered measures were administered at baseline and follow-up assessments by assessors blinded to participants' randomization status.

SECONDARY OUTCOMES:
Changes in hemoglobin A1C | Baseline assessment; 4, 8, and 12 months post-intervention assessment
  We measured participants hemoglobin A1C by means of a blood draw and laboratory test.
Changes in glucose levels | Baseline assessment; 4, 8, and 12 months post-intervention assessment
  We measured participants self-monitored glucose levels using electronic glucometers, which record the glucose level of each measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Safren, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Markowitz SM, Carper MM, Gonzalez JS, Delahanty LM, Safren SA. Cognitive-behavioral therapy for the treatment of depression and adherence in patients with type 1 diabetes: pilot data and feasibility. Prim Care Companion CNS Disord. 2012;14(2):PCC.11m01220. doi: 10.4088/PCC.11m01220. Epub 2012 Mar 15. PMID 22943030